CLINICAL TRIAL: NCT02903212
Title: Tolerance and Effectiveness of Cell Therapy by Autologous Apoptotic Cells in the Treatment of Rheumatoid Arthritis
Acronym: APO-RA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2013/196
Record Dates: First submitted 2016-09-01; First posted 2016-09-16 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Apoptotic cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rheumatoid arthritis (Experimental): Patients with rheumatoid arthritis. An injection of autologous apoptotic cells is performed on the D0.
  Interventions: Biological: Autologous apoptotic cells injection

INTERVENTIONS:
Biological: Autologous apoptotic cells injection — cells injection

SUMMARY:
The aim of the study is to determine the tolerance of apoptotic autologous cells injection in subjects with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Rheumatoid arthritis
* Therapy failure with at least one biological agent from anti-TNF-alpha (etanercept, infliximab, adalimumab, certolizumab and golimumab; 3 months at optimal dose), anti-IL6 (tocilizumab; 3 months); T-cell costimulatory pathway inhibitor (abatacept; 3 months); anti-CD20 (rituximab; 6 months at optimal dose); Anti IL-1 (anakinra; 3 months)
* Disease Activity Score (DAS) DAS28 ≥ 3.2
* Subject has provided written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Inflammatory arthritis other than rheumatoid arthritis
* History of invasive cancer
* Immunodeficiency (HIV infection, Immunosuppressive therapy)
* Active bacterial or viral infections, in particular HCV or HBV.
* Surgery not older than 4 weeks.
* Unstable comorbidities: uncontrolled diabetes, heart disease, advanced renal or hepatic impairment.
* Contraindication to an apheresis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance of apoptotic cells injection | 12 weeks
  Side effects are taken into account to assess tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Toussirot, Professor, Principal Investigator — Rhumatology - CHU Besançon

IPD SHARING:
Plan to Share IPD: No